CLINICAL TRIAL: NCT02262637
Title: Micardis® / MicardisPlus® PROTEKT (Program for Therapy Optimization With Telmisartan in Cardiovascular Diseases)
Brief Title: Micardis® / MicardisPlus® Program for Therapy Optimization With Telmisartan in Cardiovascular Diseases (PROTEKT)
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 502.441; 502.442, 502.443 (Other: Boehringer Ingelheim)
Record Dates: First submitted 2014-10-10; First posted 2014-10-13 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; telmisartan, hydrochlorothiazide drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Hypertensive patients - Cardiologists
  Interventions: Drug: Micardis®; Drug: MicardisPlus®
- Hypertensive patients - Nephrologists
  Interventions: Drug: Micardis®; Drug: MicardisPlus®
- Hypertensive patients - Diabetologists
  Interventions: Drug: Micardis®; Drug: MicardisPlus®

INTERVENTIONS:
Drug: Micardis®
Drug: MicardisPlus®

SUMMARY:
Study to evaluate efficacy and tolerability of Micardis®/MicardisPlus® under usual daily-practice prescribing-conditions with emphasis on effects on endorgan damage in the clientele of cardiologists, nephrologists, and diabetologists

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years

Exclusion Criteria:

* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients with hypertension recruited at Cardiologists, Nephrologists, Diabetologists
Sampling Method: Non-Probability Sample
Enrollment: 4814 (Actual)
Dates: Start 2003-09; Primary Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Change in systolic blood pressure (SBP) | baseline, up to 6 months
Change in diastolic blood pressure (DBP) | baseline, up to 6 months